CLINICAL TRIAL: NCT03690245
Title: Initiation of Resuscitation While Attached to the Cord With Congenital Heart Disease - INSPIRE-CHD
Brief Title: Initiation of Resuscitation While Attached to the Cord With Congenital Heart Disease
Acronym: INSPIRE-CHD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit patients
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00069732
Record Dates: First submitted 2018-09-26; First posted 2018-10-01 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-02

CONDITIONS: Congential Absence of Heart Structure; Congenital Malformation of Heart, Unspecified; Hypoplastic Left Heart Syndrome; TGA - Transposition of Great Arteries; Hypoplastic Right Heart Syndrome; Congential Malformations of Aortic Valve; Congenital Heart Defect; Congential Malformations of Great Arteries
Keywords: Congenital Heart Defect; Newborn
MeSH Terms: conditions — Heart Defects, Congenital; Hypoplastic Left Heart Syndrome; Transposition of Great Vessels

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Infants will have immediate cord clamping and respiratory support afterwards
  Interventions: Procedure: Initiation of Resuscitation While Attached to the Cord
- Initiation of Resuscitation While Attached to the Cord (Experimental): Infants will receive respiratory support for 120 seconds while attached to the cord.
  Interventions: Procedure: Initiation of Resuscitation While Attached to the Cord

INTERVENTIONS:
Procedure: Initiation of Resuscitation While Attached to the Cord — Infants will receive active resuscitative care according to the Neonatal Resuscitation Program (NRP) guidelines including warmth, dry, suctioning, oxygen, and respiratory support using iNSPiRE platform for 120 seconds while attached to the cord.

SUMMARY:
Before birth, the placenta (a structure with many blood vessels attached to the inside of your womb) and the umbilical cord (the umbilical cord is attached to the placenta) are sending oxygen and nutrients from the mother's blood through the umbilical cord to the baby. After a baby is born the cord is clamped and babies have to start breathing and support themselves.

At the moment when a baby with congenital heart disease is born they will have their cord clamped immediately (this is called immediate cord clamping (ICC)). After ICC the clinical team will start to help a baby transition by carefully monitoring their oxygen saturation (give oxygen if needed), provide warmth, and dry and stimulate. Several animal studies have shown that clamping the cord right after birth might causes the baby to miss the benefits of receiving blood from the umbilical cord / placenta.

Delayed Cord Clamping (DCC) is when the baby stays attached to the cord for a longer time. Studies show that DCC has many benefits especially for a newborn baby, such as higher iron storage, less need for blood transfusions, and improved circulation. This can be done while the baby is breathing on its own or while we help you baby breath (this is called resuscitation).

This study aims to examine whether DCC while providing resuscitation in infants with CHD is helpful compared to immediate cord clamping.

Prior to the birth of your baby, a sealed envelope will be opened and your baby will be randomly assigned to either the DCC with resuscitation group or the ICC group. 40 babies will be enrolled into this study, 20 in each group. In the DCC group, the umbilical cord will be clamped after 120 seconds during which time your baby will receive the care he/she requires by the NICU team. In the ICC group, the umbilical cord will be clamped immediately and he/she will be brought over the resuscitation bed to be cared for by the same team.

DETAILED DESCRIPTION:
Purpose: Do respiratory and cardiovascular function parameters differ in infants with congenital left heart heart disease (CHD) who receive active resuscitative care during Delayed Cord Clamping (DCC) compared to immediate cord clamping (ICC)?

Hypothesis: Infants with left heart CHD who receive active resuscitative care during DCC will have improved heart rate in the delivery room (DR) compared to those who receive ICC.

Justification: Based on our literature review, this is the first study to assess the effect of initiating resuscitation during DCC on cardiovascular function in newborn infants with left heart CHD. We speculate that initiating resuscitation during DCC will lead to a smoother transition with improving respiratory and cardiovascular stability in these infants. The results of our study will than be used to organise a large-multi-center trial.

Objectives: infants with left heart CHD who receive active resuscitative care during DCC will have improved heart rate in the delivery room (DR) compared to those who receive ICC.

Research Method/Procedures:

Study design: Randomized controlled trial.

Study population: All infants with left heart CHD born at Royal Alexandra Hospital are eligible for the study.

Intervention: Infants will be randomized to one of the following study arms:

1. Intervention group: Infants will receive active resuscitative care according to the Neonatal Resuscitation Program (NRP) guidelines including warmth, dry, suctioning, oxygen, and continuous positive airway pressure (CPAP) or PPV using iNSPiRE platform for 120 seconds during DCC.
2. Control group: Infants will have immediate cord clamping as per clinical routine.

Study protocol: Randomization: The unique trial number will be block randomized and computer generated.

Allocation Concealment: Sealed Envelope will be provided. The sealed envelopes will contain a folded card box, which allocates the unique trial number for this infant and the label "DCC group" or "ICC group".

Blinding: There will be no blinding, as it would not be feasible to conduct resuscitation without the resuscitation team knowing the actual intervention that the subject will receive.

Intervention group: The infant will be placed on iNSPiRE platform, the airway will be cleared if necessary; the baby will be dried and stimulated, and pulse oximeter will be placed on the right wrist. CPAP will be administered using T-piece resuscitator at 6 cmH2O, with FiO2 of 21%. PPV will be provided at an initial peak inspiratory pressure (PIP) of 24 cmH2O and rate of 40-60 bpm in case of apnea, gasping breathing or heart rate <100 bpm. Interventions will be recorded at 10 seconds intervals; while vital signs will be recorded at 30 seconds intervals. At 120 seconds after birth, the cord will be clamped and the platform will be wheeled to the radiant warmer in the delivery room, the baby will be transferred on CPAP, and resuscitation/transitional care will continue according to the institutional guidelines. If immediate intubation or chest compressions are required despite initiating CPAP or PPV via mask and T-piece resuscitator, the procedure will be interrupted, the cord will be clamped, and the baby transferred to the radiant warmer.

Control group: Infants randomized to the control arm will have immediate cord clamping as per hospital guidelines. Once on the radiant warmer, airway will be cleared, and pulse oximeter placed on the right wrist and routine resuscitation care as per hospital guidelines.

Management in the delivery room on the radiant warmer for all study groups: The subsequent management of the infant in the delivery room will follow the institutional guidelines. In addition, we will use Philips NM3 Respiratory Function Monitor (RFM), placed on a special trolley/platform to measure the delivered airway pressures, tidal volume (VT), and ECO2 using a flow sensor placed between the face mask (or the endotracheal tube in case of intubated infant) and the T-piece resuscitator. The pulse oximeter sensor will be connected to the RFM. The RFM display screen will show only the SpO2, and other parameters will be concealed from the resuscitation team. The RFM will be connected to a laptop to allow real time data acquisition. A video camera mounted on the top of the radiant warmer will be used to record the management and will stream to the same laptop. Axillary temperature will be measured once the infant is transferred to the radiant warmer and at 10 minutes of age. Once the infant is stable he/she will be transferred to the NICU.

Management in the NICU: Infants will be managed according to the institutional guidelines. Neonatal Echocardiography will be performed at 6 and 24 hours of age to assess cardiac function.

Plan for data analysis:

Pregnancies complicated by fetal left heart CHD will be recruited through the Fetal & Neonatal Cardiology Program at the Royal Alexandra Hospital over a period of 24 months. Approximately another three months will be required to collect hospital data on all infants enrolled. Resuscitation data will be collected on a standard form (Neonatal Resuscitation Record) that will form part of each infant's hospital record. Other medical data on each infant will be collected on Case Report Forms and hemodynamic data will be generated in the first 24 hours as part of the routine care of these infants on the David Schiff NICU.

The signals of airway flow, tidal volume, airway pressure, and exhaled CO2 will be recorded at 200Hz using Spectra physiological recording program (a customized neonatal respiratory physiology program). A breath-by-breath analysis will be performed manually for the duration of each recording. Tidal volume, inflation time, gas flow and exhaled CO2 will be measured.

Descriptive statistics will be used to describe the population. We will use student t-test, Mann Whitney U test for continuous variables and Chi square test or Fisher Exact Test for categorical variables to compare the groups as appropriate. Randomized infants will be analyzed in their respective groups regardless of the actual intervention received following the intension-to-treat concept. However, a priori subgroup comparison will be performed between the following groups:

1. Infants randomized to resuscitative care for 120 seconds.
2. Infants randomized to the control group.

Sample size: This is a feasibility trial and we estimate to recruit 40 infants (20 per group) to assess feasibility of this approach.

ELIGIBILITY:
Inclusion Criteria:

* Infants with rights or left heart congenital malformation

Exclusion Criteria:

* Infants with no heart congenital malformation

Max Age: 20 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Increase in heart rate | At 5 minutes after birth

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No